CLINICAL TRIAL: NCT06619730
Title: Using Brain Function Monitors to Guide Anesthetic Management in Improving Anesthesia Recovery: a Randomized Pilot Study to Compare Outcomes in Young Adult Patients.
Brief Title: Brain Function Monitoring During Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB24-0454
Record Dates: First submitted 2024-08-07; First posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Surgery
Keywords: Brain function Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Arm (No Intervention): Conventional method: Anesthesia will not be guided by the Sedline brain function monitor during the procedure.
- Sedline Monitor Arm (Active Comparator): Anesthesia care guided by Sedline brain function monitor during the procedure.
  Interventions: Device: Sedline Brain Function Monitor

INTERVENTIONS:
Device: Sedline Brain Function Monitor — The anesthesia provider will use the Sedline Brain Function Monitor information to affect their anesthetic dosing.
  Arms: Sedline Monitor Arm

SUMMARY:
The purpose of this research is to gather information on the effectiveness of the Sedline Brain Function Monitor, and its use in this study to determine whether monitoring the brain activity during anesthesia will improve recovery, including earlier discharge and less side effects. Furthermore, the study team wants to determine whether males and females respond to anesthetics in a similar manner with and without brain monitoring.

DETAILED DESCRIPTION:
Screening: One day prior to surgery or the day-of surgery in the preoperative holding area Once potentially appropriate subjects have been identified from the OR schedule for the next day, the study team will contact the anesthesia provider (resident, nurse aestheticist, attending) who is scheduled to treat that patient and explain to him/her about the research project and ask them to use a Sedline Brain Function Monitor for the case. In explaining the research project to anesthesia providers, the study team will stress the importance of keeping the patient's Sedline Density Spectral Array (DSA) between 8-15 or/and Patient State Index (PSI) reading between 25-50 throughout the course of the case in the subjects who are randomly selected in the monitoring group. If the blood pressure (BP) or heart rate (HR) is over 25-30 % baseline, an opioid or other pain medications will be used first, before increasing the dose of inhalational agent or propofol. If BP is low and PSI is on the low end, study team will lower the inhalational agent or propofol first. If the patient moves and BP and PSI are within the ranges, muscle relaxant may be given first unless the use of muscle relaxant is not allowed for the surgical reason. If both opioids and muscle relaxant adjustment fail to achieve the hemodynamic stability and immobility goal, then the study team will adjust the doses of inhalational agent or propofol.

Treatment: During general anesthesia for surgery projected to last 60-240 mins The study team will try to treat the need of each component in general anesthesia, unconsciousness, immobility, nociception and hemodynamic stability accordingly while the study team understands the 4 components are interlinked. In the non-monitoring group (control or conventional group), the anesthesia providers will administer the anesthetics in the conventional manner, mainly based on the hemodynamic responses and the minimum alveolar concentration (MAC) of inhalational agents during the surgery. The brain activities are not usually monitored in real time by a brain monitor. The anesthesia providers are allowed to use inhalational, intravenous anesthetic agents, opioids and muscle relaxants to produce adequate general anesthesia in both groups. Overall anesthesia care during the surgery will not be compromised.

On the day of planned surgery, the study team will meet with each patient in pre-op and ask for their informed consent to participate in this research. If they agree to participate, their anesthesia provider will apply a Sedline Monitor to their forehead during the general anesthesia procedure. The anesthesia provider may use the data from the monitor to affect their anesthetic administration, or may cover the data from the monitor and only use conventional measures to guide anesthetic dosing in these control cases (blood pressure, heart rate, body movement, respiratory rate, MAC of inhalational agent), depending on what group into which the patient has been randomized.

Once the general anesthesia procedure is over and the patient is recovering in pediatric acute care unit (PACU), the study team will meet with each patient again, and use a standardized survey to ask about their satisfaction with their anesthetic, including questions about their post-operative pain and feelings of nausea or presence of vomiting.

Follow-up: Follow up on postoperative day 1 via phone call The study team will follow-up with each patient via phone call on post-op Day 1 and ask the same survey questions to ensure resolution of their symptoms and timing of the resolution of their symptoms. The study time will also ask the PACU nurse to record at what time the patient met the University of Chicago Medical Center (UCMC)-specific PACU discharge protocol criteria.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Physical Status Classification Grade of 1(normal, healthy patient) to Grade 3 (patient with severe disease)
* Between ages 18-45 years old
* Planned surgery duration between 60-240 minutes General-endotracheal-tube-anesthesia or general anesthesia with laryngeal mask airway
* Subjects capable of giving informed consent or
* Subjects who have an acceptable surrogate capable of giving consent on behalf of the subject
* All contraception methods will be allowable for any subject in this study. Participants may opt-out of a pregnancy test if they would prefer to proceed with surgery without one.

Pregnant women will not be strictly excluded from this study if they meet all other criteria.

Exclusion Criteria:

* American Society of Anesthesiology Physical Status Classification Grade of 4,5,6 (diseases that are life threatening or no possibility of survival)
* Listed allergies to any commonly used anesthetic agents
* History of seizures, as a seizure while using brain monitoring may influence the anesthesia provider in a way that is not aligned with the purpose of this study
* Any patient undergoing emergency surgery, as can not be ensured that consent will be able to be properly obtained
* Patient refusal to participate in study
* Any patient undergoing surgery that would prevent placement of the Sedline monitor leads (for example - surgery on the patient's forehead/scalp)
* Patients who receive neuraxial anesthesia or a peripheral nerve block as part of their anesthetic
* Patients who are taking gender-affirming hormonal medications, as this can affect the response to anesthetics
* The duration of surgery scheduled <60 minutes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Speed of recovery time | Up to 3 hours
  The primary endpoint is the speed of recovery time, measured from the end time of the surgery, to the time of meeting the criteria for pediatric acute care unit (PACU) discharge. These criteria are lack of nausea/vomiting, grogginess and the level of pain; with 1 being no pain and 10 being severe pain.

SECONDARY OUTCOMES:
To assess patient satisfaction with their anesthetic experience and side effects. | Up to 1 day post surgery
  This will be done via a post-op survey, that measures pain levels, as before, and if the patient is experiencing any residual ill effects.
Difference in recovery times between males and females | Up to 2 days post surgery
  To determine if the use of the Sedline Brain Function Monitor will affect the recovery time differently between males and females. Differences may be attributed to the differences in brain waves.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Xie, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States